CLINICAL TRIAL: NCT00656461
Title: Phase 1 Study of MKC-1 in Patients With Advanced or Metastatic Solid Malignancies
Brief Title: Phase 1 Study of MKC-1 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Chief Medical Officer, Miikana Therapeutics, an EntreMed, Inc. company
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC-106
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Advanced Cancer
Keywords: Advanced cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MKC-1

INTERVENTIONS:
Drug: MKC-1 — 30 mg and 100 mg capsules, dosed BID daily on a continuous schedule

SUMMARY:
This is an open-label study to determine the highest dose of MKC-1 that may be administered daily on a continuous basis for patients with advanced or refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative measures do not exist or are no longer effective.
* Age greater than or equal to 18 years.
* ECOG performance status ≤1
* ANC greater than or equal to 1,500/mm3;
* Platelets greater than or equal to 100,000/mm3
* creatinine ≤1.5 times institutional upper limit of normal (ULN)
* T Bili within normal limits;
* AST and ALT less than or equal to 2.5 times ULN; and
* albumin greater than or equal to 3.0 g/dL
* have measurable disease by RECIST, radiographically evaluable disease, or detectable disease
* women of child-bearing potential and men must agree to use adequate contraception
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Have previously received MKC-1.
* Have received radiation to greater than 25% of the bone marrow.
* Have had anti-cancer therapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Are concurrently receiving any other investigational agents while on study.
* Have known brain metastases
* Have any condition that impairs the ability to swallow and retain MKC-1 capsules.
* Uncontrolled intercurrent illness
* Are pregnant or breastfeeding
* HIV-positive patients
* Patients with uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of MKC-1 administered orally twice a day (bid) continuously in patients with advanced or refractory solid tumors. | Throughout study participation

SECONDARY OUTCOMES:
Determine evidence of benefit in cancer patients when MKC-1 is administered orally twice a day (bid) continuously by evaluating tumor response and/or tumor marker improvement. | During study participation

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Liu, MD, Principal Investigator — U. of Wisconsin
Locations (1):
- U. of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin, United States